CLINICAL TRIAL: NCT02006927
Title: A Pilot Study of the Feasibility of Chronic Cavernous Nerve Stimulation to Promote Neural Regeneration and Erectile Function
Brief Title: A Pilot Study of the Feasibility of Chronic Cavernous Nerve Stimulation to Promote Regeneration and Erectile Function
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of Enrollment
Sponsor: Kenneth M Peters, MD (Other)
Collaborators: Corewell Health East (Other)
Responsible Party: Sponsor-Investigator, Kenneth M Peters, MD, Chief of Urology, Corewell Health East
Organization: Corewell Health East (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-420
Record Dates: First submitted 2013-12-04; First posted 2013-12-10 (Estimated); Results first posted 2020-10-01 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Nerve Stimulation (Experimental): Placement and stimulation of implantable neurostimulation device/leads post radical robotic prostatectomy
  Interventions: Device: Nerve Stimulation

INTERVENTIONS:
Device: Nerve Stimulation — Placement and stimulation of implantable neurostimulation device/leads post radical robotic prostatectomy
  Other Names: Lead stimulation

SUMMARY:
The goal of this study is to evaluate electrical stimulation of nerves responsible for erectile function after surgery to remove the prostate (prostatectomy). Electrical stimulation of the nerves responsible for erectile function is experimental. The investigators hypothesize that the subjects can tolerate nerve stimulation.

DETAILED DESCRIPTION:
The objective of the study is to explore the feasibility of using an implantable neurostimulation device/leads post radical robotic prostatectomy as a method for enhancing neural recovery/penile rehabilitation and/or erectile dysfunction treatment. This will be a single center pilot study of up to 10 patients. The leads will be placed and stimulated intraoperatively to assess proper placement and stimulation parameters needed to achieve change in penile length and/or circumference. One week post operatively, the leads will be connected to an external stimulator device and activated. Subjects will be instructed to stimulate each lead by turning on the device each day for up to six weeks. The leads will be removed at six weeks post operative and subjects will be followed for up to two years.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled for a robotic radical prostatectomy procedure with bilateral nerve sparing.
2. Sexually functional preoperatively as defined by a Sexual Health Inventory For Men (SHIM) score of greater than 21 at baseline off any phosphodiesterase 5 inhibitors.
3. Without erectile dysfunction treatment in the 12 months prior to radical prostatectomy.
4. Willing to stop phosphodiesterase 5 inhibitor that has only been started prophylactically to promote penile rehabilitation after prostatectomy.
5. Age 40 to 80 years of age.
6. Stable on all medications for at least 6 weeks prior to completing baseline measures and be willing to remain on those medications with no dose adjustments expected for 6 weeks post-implantation.
7. An appropriate candidate for the surgical procedure required for this study.
8. Willing and able to comply with all study related procedures and visits, and making accurate daily entries into a diary for approximately 6 weeks post radical prostatectomy (lead stimulation phase).
9. Capable of reading and understanding patient information materials and giving written informed consent.

Exclusion Criteria:

1. Have been diagnosed with vascular insufficiency to any pelvic blood vessels.
2. Have prior surgical implantation of penile prosthesis, or other prior major pelvic surgery.
3. History of significant pelvic trauma.
4. Are current substance abusers including illicit drugs or use narcotics more than 15 days/month.
5. Have a significant psychiatric disorder or under current treatment with antipsychotic or antidepressive medications.
6. Have previously not tolerated an implanted medical device and subsequently required explant of the device for any reason other than device malfunction.
7. Have a condition currently requiring or likely to require the use of MRI or diathermy.
8. Currently have an active implantable device.
9. Have participated in any drug or device trial in the last 4 weeks or plan to participate in any other drug or device study during the next 24 months.
10. Have metabolic or immunodeficiency disorders related to recurrent infections, specifically including but not limited to diabetes mellitus, HIV, disorders requiring chronic or high dose corticosteroids, or connective tissue disorders.
11. Have Peyronies disease.
12. Subject possesses any other characteristics that, per the investigator's judgment, deems them unsuitable (eg increases risk, impairs data collection, etc) for the procedure/study.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M Peters, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nerve Stimulation
Started | 3
Completed | 0
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Baseline data was collected on all 3 participants before they withdrew from study
Arm/Group | Nerve Stimulation
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Tolerability of Nerve Stimulation
Description: Evaluate the safety and tolerability of chronic cavernous nerve stimulation post radical prostatectomy by measuring the incidence of major complications that may include lead removal, infection at the site or painful stimulation requiring lead removal.
Time Frame: 6 weeks
Population: All participants withdrawn from study prior to any data collection or analysis. No data analyzed to report.
Arm/Group | Nerve Stimulation
Number analyzed (Participants) | 0

2. Secondary Outcome: Efficacy of Nerve Stimulation
Description: Explore the potential efficacy of chronic cavernous nerve stimulation on the return of erectile function post radical prostatectomy. Measures to assess efficacy include direct response to stimulation, changes in penile tumescence (girth) and sensory perception.
Time Frame: 24 months
Population: All participants withdrawn from study prior to any data collection or analysis. No data analyzed to report.
Arm/Group | Nerve Stimulation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 24 months
Description: Adverse events (AEs) assessment will be performed at each study visit following implantation through 24 months. All AEs will be initially reviewed by the Principal Investigator (PI), The PI will determine severity and causality. AEs will be reported per institutional and FDA requirements.
Arm/Group | Nerve Stimulation
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nerve Stimulation (N=3)
Nausea/vomiting (Gastrointestinal disorders) | 1 (1)
Device lead migration (Reproductive system and breast disorders) | 3 (3)
Hematuria (Renal and urinary disorders) | 2 (2)
Infected pelvic hematoma (Reproductive system and breast disorders) | 2 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bladder leak (Renal and urinary disorders) | 1 (1)
Hiatal hernia (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated early after technical problems with device caused device removal in all 3 enrolled subjects and withdrawal of all 3 enrolled subjects prior to data collection or analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes